CLINICAL TRIAL: NCT05526066
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Nested Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ARCT-810 in Adolescent and Adult Participants With Ornithine Transcarbamylase Deficiency
Brief Title: Study for Adolescents and Adults With Ornithine Transcarbamylase Deficiency to Evaluate Safety and Tolerability of ARCT-810
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after the completion of Cohort 1 (0.3 mg/kg) due to slow enrollment in this placebo-controlled study.
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARCT-810-03
Record Dates: First submitted 2022-08-08; First posted 2022-09-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Ornithine Transcarbamylase Deficiency; OTC Deficiency; OTCD
Keywords: OTC; OTCD; Ornithine; Transcarbamylase; mRNA; Ornithine Transcarbamylase Deficiency; OTC Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Intervention Model Description: On Day 1, participants will receive a single dose of Study Drug via intravenous infusion.
  If the safety observations are considered acceptable, that participant will enter the multiple-dose portion of the study in which they will receive a further 5 doses of Study Drug on Days 15, 29, 43, 57 and 71.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARCT-810 (Experimental): Participants receive an initial intravenous (IV) infusion ARCT-810. If considered safe and well tolerated, participants will receive up to 5 additional IV infusions of ARCT-810 administered at 14-day intervals.
  Interventions: Biological: ARCT-810
- Placebo, Normal Saline (Placebo Comparator): Participants receive an initial IV infusion of placebo. If considered safe and well tolerated, participants receive up to 5 additional IV infusions of placebo administered at 14-day intervals.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARCT-810 — ARCT-810 is messenger RNA (mRNA) coding for Ornithine Transcarbamylase (OTC) formulated in a lipid nanoparticle (LNP).
  Arms: ARCT-810
Other: Placebo — Normal Saline
  Arms: Placebo, Normal Saline

SUMMARY:
The primary objective is to evaluate the safety and tolerability of repeated doses of intravenously administered ARCT-810.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, placebo-controlled study of ARCT-810 in people living with OTC deficiency 12 years of age and older. After an at least 4 week screening and diet stabilization period, participants will be randomized 3:1 to receive ARCT-810 or placebo. Following the first dose and safety evaluation, participants will receive up to an additional 5 doses of ARCT-810 or placebo, each separated by 14 days. The treatment period is followed by a 12-week observation period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adequate cognitive ability to understand study requirements and give informed consent
2. Males and females aged 12 to 65 years inclusive, at Screening
3. Documented diagnosis of OTC deficiency
4. Clinical stability (no clinical symptoms of hyperammonemia within 1 month, no hospitalizations for metabolic decompensation within 3 months, ≤ 2 hospitalizations within 1 year)
5. Stable protein-restricted diet, dietary supplements, and ammonia scavenger regimen (if applicable) for at least 28 days.
6. BMI = 18.0 - 32.0 kg/m2, inclusive for adults, and >5th percentile for adolescents ≥12 to 17 years
7. Must be willing to adhere to contraception guidelines

Key Exclusion Criteria:

1. History of any OTC gene therapy, or history of liver-derived stem cell therapy in the past 3 years
2. History of other medical conditions that may make the participant unsuitable for inclusion or could interfere with study participation (e.g., uncontrolled hypertension or diabetes, malignancy, HIV, hepatitis B or C)
3. History of severe allergic reaction to liposomal or PEG-containing products
4. Abuse of illicit drugs, medications or alcohol
5. Clinically significant laboratory abnormalities on screening labs

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of adverse events (AEs) | Week 23
  Safety and tolerability of ARCT-810 assessed by determining the number and severity of AEs by dose level

SECONDARY OUTCOMES:
Plasma concentration area under the curve after first and last doses of ARCT-810 | Up to 17 Weeks
  Area under the plasma concentration versus time curve (AUC) from time zero to the last quantifiable time point
Maximum observed plasma concentration (Cmax) after first and last doses of ARCT-810 | Up to 17 Weeks
  The maximum observed plasma concentration (Cmax)
Time at which Cmax occurred after first and last doses of ARCT-810 | Up to 17 Weeks
  The time at which Cmax occurred (Tmax)
AUC0-inf after first and last doses of ARCT-810 | Up to 17 Weeks
  Plasma AUC from time zero extrapolated to infinity
AUCExtrap after first and last doses of ARCT-810 | Up to 17 Weeks
  The relative portion of AUC0-inf extrapolated beyond AUC0-t
T1/2 after first and last doses of ARCT-810 | Up to 17 Weeks
  Terminal half-life
MRT0-inf after first and last doses of ARCT-810 | Up to 17 Weeks
  The mean residence time extrapolated to infinity
CL after first and last doses of ARCT-810 | Up to 17 Weeks
  Total body clearance, calculated as dose divided by AUC0-inf
Vss after first and last doses of ARCT-810 | Up to 17 Weeks
  Volume of distribution
Urea Cycle Function | Week 12
  Change from baseline in urea cycle function as measured by 13C-urea assay
Plasma Ammonia | Week 11
  Change from baseline in urea cycle function as measured by 24-hour plasma ammonia profile

CONTACTS AND LOCATIONS:
Locations (14):
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- France (2):
  - Hôpitaux Universitaires de Marseille - Hôpital de la Timone, Marseille
  - Assistance Publique - Hôpitaux de Paris (AP-HP) - Hôpital Necker-Enfants Malades, Paris
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Ospedale Pediatrico Bambino Gesu, Rome
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario Universitario de Santiago (CHUS) - Hospital Clínico Universitario, Santiago de Compostela
- Karolinska Universitetssjukhuset - Astrid Lindgrens Barnsjukhus, Stockholm, Sweden
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust - Queen Elizabeth Hospital Birmingham, Birmingham, UK
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London, UK
  - University College London Hospitals NHS Foundation Trust - National Hospital for Neurology and Neurosurgery, London
  - Salford Royal NHS Foundation Trust - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No